CLINICAL TRIAL: NCT01684384
Title: Correlation of Functional Respiratory Imaging Parameters With Lung Function Parameters and Patient Reported Outcome Measures During Exacerbation of COPD.
Brief Title: Research to Evaluate a Possible Relation Between Values Obtained After Processing CT Images, Lung Function Tests and the Experience of the Patient During an Exacerbation in COPD Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLUI-2011-79
Record Dates: First submitted 2012-09-06; First posted 2012-09-13 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; COPD; Exacerbation; Functional Respiratory Imaging; High Resolution Computed Tomography; HRCT scan; Patient Reported Outcome; PRO; Computational Fluid Dynamic; CFD; Lung function parameters
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No treatment (Experimental): CT-scans will be taken in the study. The EC of the University hospital antwerp considers this as an intervention.
  Interventions: Radiation: Functional Respiratory Imaging

INTERVENTIONS:
Radiation: Functional Respiratory Imaging — HRCT scan at FRC and TLC as taken during an episode of exacerbation and after recovering.
  Other Names: HRCT scan

SUMMARY:
In this study the consequences of exacerbations will be visualized by high resolution computed tomography (HRCT) scan at functional residual capacity (FRC) and total lung capacity (TLC) as taken during an episode of exacerbation and after recovering. Changes in HRCT based airway dimensions and computational fluid dynamic (CFD) -based resistance values will be correlated with changes in patient reported outcomes (PROs) and lung function tests recorded at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 40 years old
* COPD as defined by the global Initiative on obstructive lung disease4
* Post-bronchodilator FEV1/FVC < 70% AND post-bronchodilator FEV1 <80%pred as documented in the last 5 years.
* Smoking history of at least 10 pack-years
* At entry in the study experiencing an exacerbation defined as an acute change in the patient 's baseline dyspnea, cough, and/or sputum that is beyond normal day to day variations, and that necessitates the administration or doubling of systemic corticosteroid treatment.
* Patients must be able to understand and complete protocol requirements, instructions, questionnaires and protocol-stated restrictions.
* Written and signed informed consent

Exclusion Criteria:

* Pregnant or lactating females
* Patient diagnosed with asthma
* Patient with pneumonia as defined radiologically at the start of the exacerbation
* Patient with a history of or presence of lung cancer
* Patient with an indication for non-invasive ventilation
* Patient unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study.
* Patient who received any investigational new drug within the last 4 weeks prior to visit 1.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Changes in functional respiratory imaging parameters | Baseline (= during exacerbation) and after about 6 weeks (= after recovering)
  The primary objective of this study is to evaluate whether changes in HRCT based airway dimensions and Computational Fluid Dynamic (CFD)-based resistance values correlate with changes in lung function parameters, under the conditions of exacerbation of COPD as well as after recovering from exacerbation.
Changes in lung function parameters | Baseline (= during exacerbation) and after about 6 weeks (= after recovering)
  The primary objective of this study is to evaluate whether changes in HRCT based airway dimensions and Computational Fluid Dynamic (CFD)-based resistance values correlate with changes in lung function parameters, under the conditions of exacerbation of COPD as well as after recovering from exacerbation.

SECONDARY OUTCOMES:
Changes in patient reported outcome (PRO) measures | Baseline (= during exacerbation) and after about 6 weeks (= after recovering)
  The secondary objective is to check if the changes in CFD data actually correlate better with changes in PRO than changes in lung function parameters.

OTHER OUTCOMES:
Reproducibility of segmentation | Within 1 month of visit
  As tertiary objective the reproducibility of the segmentations done by the centers will be evaluated. To accomplish reproducible segmentations the multiple centers will be guided to perform accurate segmentations, and bottlenecks in the usage of the program will be identified and resolved in order to simplify it where necessary and possible.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp; Huib AM Kerstjens, MD, Principal Investigator — University Medical Center Groningen; Emiel FM Wouters, MD, Principal Investigator — Maastricht University Medical Center; Massimo Pistolesi, MD, Principal Investigator — University of Florence
Locations (4):
- Antwerp University Hospital, Edegem, Antwerp, Belgium
- University of Florence, Florence, Italy
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Maastricht University Medical Center, Maastricht